CLINICAL TRIAL: NCT00635180
Title: Changes in Intraocular Pressure and Pulsatile Ocular Blood Flow Measured Continuously During Isometric Exercise
Brief Title: Intraocular Pressure (IOP) and Isometric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Sven Ove Semb, MD PhD, Ullevål University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UUS-IOP-07
Record Dates: First submitted 2008-02-05; First posted 2008-03-13 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-02

CONDITIONS: Intraocular Pressure
Keywords: Isometric exercise; intraocular pressure; Physiological changes in intraocular pressure during isometric exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 1: Healthy subjects
  Interventions: Behavioral: isometric exercise

INTERVENTIONS:
Behavioral: isometric exercise

SUMMARY:
The purpose of this study is to investigate changes in intraocular pressure measured continuously during isometric exercise.

ELIGIBILITY:
Inclusion Criteria:

* Young, healthy subjects

Exclusion Criteria:

* Known ocular diseases
* Previous ocular trauma

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven O Semb, MD, PhD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Eye dpt, Ullevaal University Hospital, Oslo, Oslo County, Norway